CLINICAL TRIAL: NCT07188506
Title: Youth Suicide Risk Factors: Clinical, Neuroimaging, Genetic, and Microbiome Insights, and Predictors of Response to Deep Transcranial Magnetic Stimulation (dTMS)
Brief Title: Youth Suicide Risk Factors, Reduction of Suicide Risk Factor in Youth People
Acronym: YOU-SURF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 8012
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Mood Disorders; Suicide, Attempted; Suicidal Ideation; Suicide Prevention
MeSH Terms: conditions — Mood Disorders; Suicide, Attempted; Suicidal Ideation; Suicide Prevention | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Suicidal clinic group (Experimental): 60 patients at suicidal risk
  Interventions: Diagnostic Test: Clinical and blood parameters; Genetic: Illumina Infinium Global Screening Array 4.0 (GSA 4.0); Device: dTMS treatment
- Not-Suicidal clinic group (Experimental): 60 patients without suicidal risk
  Interventions: Diagnostic Test: Clinical and blood parameters; Genetic: Illumina Infinium Global Screening Array 4.0 (GSA 4.0); Device: dTMS treatment
- Healthy Controls (Active Comparator): 60 healthy controls (HCs)
  Interventions: Diagnostic Test: Clinical and blood parameters; Genetic: Illumina Infinium Global Screening Array 4.0 (GSA 4.0)

INTERVENTIONS:
Diagnostic Test: Clinical and blood parameters — Clinical data and MRI measurements
  Other Names: Magnetic Resonance Imaging (MRI) protocol
Genetic: Illumina Infinium Global Screening Array 4.0 (GSA 4.0) — Genomic analyses
  Other Names: Microbiota protocol
Device: dTMS treatment — high-intensity deep transcranial magnetic stimulation (dTMS) device recognized for clinical application in mood disorders
  Arms: Not-Suicidal clinic group; Suicidal clinic group

SUMMARY:
The YOU-SURF project is at the forefront of youth suicide prevention, with the goal of integrating multimodal clinical and neurobiological data to comprehensively identify risk factors and the most effective intervention strategies. Suicide is one of the leading causes of death among young people, with particularly alarming incidence rates during adolescence and early adulthood. Suicidal risk is a complex phenomenon, determined by a multiplicity of clinical, environmental, and biological factors. Emerging evidence suggests that information derived from neuroimaging, genetics, and the microbiome may also play a significant role. However, studies conducted to date have not yet adopted a truly multimodal approach that jointly integrates these dimensions in the identification of risk factors for suicide in youth. The YOU-SURF project aims to fill this critical gap.

YOU-SURF will also pioneer the use of deep transcranial magnetic stimulation (dTMS), an innovative neuromodulation technique, whose effectiveness in reducing suicidal risk in young people will be assessed within a longitudinal design. Although some preliminary evidence suggests a potential benefit of neuromodulation treatments in this population, the specific effects of dTMS on suicidal risk in youth remain largely unexplored. Furthermore, there is a significant lack of knowledge regarding predictors of response to dTMS in young individuals at risk for self-harming behaviors.

The specific objectives of the project are as follows:

1. To identify youth suicide risk factors through the integration of clinical, environmental, neuroimaging, genetic, and microbiome data;
2. To longitudinally evaluate the effectiveness of dTMS in the treatment of young people at risk of suicide;
3. To develop a predictive model based on machine learning techniques, grounded in multimodal data, to estimate the individual response to dTMS in this population.

The results of the project will provide a solid scientific basis for the development of personalized prevention and treatment interventions, improving clinical effectiveness and resource allocation in youth mental health services.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mood disorder (major depressive episode, major depressive disorder, or bipolar disorder) according to DSM-5;
* Age between 18 and 25 years;
* Eligibility for magnetic resonance imaging;
* Proficiency in the Italian language.

Exclusion Criteria:

* Comorbidity with severe neurological or medical conditions;
* Diagnosis of cognitive impairment;
* Inability to provide informed consent.

For the control group:

Inclusion Criteria:

the same as the experimental group.

Exclusion Criteria:

* subjects with DSM-5 disorders
* subjects with a family history of psychiatric disorders will be excluded.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Change of suicidal risk | 3 months
  Reduction of suicidal risk, assessed using the Columbia Suicide Severity Rating Scale (C-SSRS) score (No, Low, Moderate, High)

SECONDARY OUTCOMES:
Severity of depressive symptoms | 3 months
  Severity of depressive symptoms, assessed with the Montgomery-Åsberg Depression Rating Scale (MADRS):
  0 to 6: normal/symptom absent 7 to 19: mild depression 20 to 34: moderate depression 35 to 60: severe depression
General psychiatric symptoms | 3 months
  General psychiatric symptoms measured with the Brief Psychiatric Rating Scale (BPRS).
  The rater enters a number for each symptom construct that ranges from 1 (not present) to 7 (extremely severe).

CONTACTS AND LOCATIONS:
Overall Officials: Delfina Janiri, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS - UOC Psichiatria Clinica e d'Urgenza, Roma, RM, Italy